CLINICAL TRIAL: NCT02951390
Title: High Definition White-Light Colonoscopy Versus Chromoendoscopy for Surveillance of Lynch Syndrome. A Prospective, Multicenter and Randomized Study
Brief Title: High Definition White-Light Colonoscopy vs. Chromoendoscopy for Surveillance of Lynch Syndrome.
Acronym: EndoLynch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, María Pellisé, MD. PhD. Consultant, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2016/0440
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Lynch Syndrome
Keywords: Surveillance; Colorectal cancer; Colonoscopy; Adenoma; Chromoendoscopy
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-definition white-light endoscopy (Active Comparator): High-definition white-light endoscopy without indigo carmine instilation
  Interventions: Other: High-definition white-light endoscopy
- High-definition chromoendoscopy (No Intervention): High-definition indigo-carmine chromoendoscopy

INTERVENTIONS:
Other: High-definition white-light endoscopy — The intervention is do not perform chromoendoscopy
  Arms: High-definition white-light endoscopy

SUMMARY:
Adenomas in Lynch syndrome have an accelerated progression to colorectal cancer (CRC) which might occur despite a regular follow-up. Despite low evidence, high-definition technology (HD) and indigo-carmine chromoendoscopy (CE) are recommended for surveillance in Lynch syndrome.The investigators will conduct a prospective multicenter randomized non-inferiority study. The principal aim is to compare the adenoma detection rate with WLE vs CE. Our hypothesis is that HD-white-light endoscopy (WLE) is not inferior to CE. Therefore - under expert hands - HD-CE does not add any significant advantage over HD-WLE on adenoma detection rate in patients with Lynch syndrome.

DETAILED DESCRIPTION:
The investigators will conduct a prospective multicenter randomized non-inferiority study. Eligible patients will be those with Lynch syndrome (known germline mutation in mismatch repair genes) who undergo surveillance colonoscopies. Patients will be sequentially assigned in a 1:1 ratio to HD-WLE or HD-CE. The method of stratified randomization based on partial colectomy history will be used to avoid proportion imbalance between groups. Participant centers must have an organized high-risk of CRC clinic and endoscopic unit provided with HD technology. Endoscopists must have a documented high adenoma detection rate and experience in performing CE in patients with high-risk conditions of CRC.

The principal aim is to compare the adenoma detection rate with WLE vs CE. Principal outcome measures will be: 1) adenoma detection rate, defined as the proportion of patients with at least one adenoma in each arm; 2) number of adenomas per patient, defined as the total number of detected adenomas in each arm (HD-WLE or HD-CE) divided by the number of colonoscopies in each arm.

The sample size calculation was determined for a non-inferiority study. Assuming an ADR of 28% with conventional chromoendoscopy in patients with Lynch syndrome, a 15% non-inferiority margin, a one-sided significance level of 0.05 powered at 80% and a 10% of drop-off. Based on these assumptions, it was determined that 122 patients were required for each arm (a total of 244).

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven pathologic germline mutation in one of the mismatch-repair (MMR) gene (MLH1, MSH2, MSH6, PMS2 or Epcam) who will undergo surveillance colonoscopy

Exclusion Criteria:

* Patients with total colectomy
* Concomitant inflammatory bowel disease
* Inadequate bowel preparation (Boston scale <2 in any colonic segment)
* Incomplete procedure (without intubation of cecum or ileo-colonic anastomosis)
* Previous colonoscopy in less than one year
* Inability to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | one year
  Adenoma detection rate is defined as the proportion of patients with at least one adenoma in each arm

SECONDARY OUTCOMES:
Mean of adenomas per patient | one year
  the total number of adenomas detected in each group (HD-WLE or HD-CE) divided by the number of colonoscopies in each group
Mean number per patient of total polyps | one year
Mean number per patient of total serrated lesions | one year
Polyp detection rate | one year
Serrated lesions detection rate | one year
Withdrawal time | 30 minutes
  Extubation time from the cecum to scope removal from the anus, with exception of time taken for any therapeutic intervention
Total procedure time | 30 minutes
  Starting with endoscope insertion and withdrawal time including therapeutic interventions

CONTACTS AND LOCATIONS:
Overall Officials: María Pellisé, MD. PhD., Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- María Pellisé. MD. PhD., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurlstone DP, Karajeh M, Cross SS, McAlindon ME, Brown S, Hunter MD, Sanders DS. The role of high-magnification-chromoscopic colonoscopy in hereditary nonpolyposis colorectal cancer screening: a prospective "back-to-back" endoscopic study. Am J Gastroenterol. 2005 Oct;100(10):2167-73. doi: 10.1111/j.1572-0241.2005.41481.x. PMID 16181364
- [Background] Lecomte T, Cellier C, Meatchi T, Barbier JP, Cugnenc PH, Jian R, Laurent-Puig P, Landi B. Chromoendoscopic colonoscopy for detecting preneoplastic lesions in hereditary nonpolyposis colorectal cancer syndrome. Clin Gastroenterol Hepatol. 2005 Sep;3(9):897-902. doi: 10.1016/s1542-3565(05)00403-9. PMID 16234028
- [Background] Stoffel EM, Turgeon DK, Stockwell DH, Zhao L, Normolle DP, Tuck MK, Bresalier RS, Marcon NE, Baron JA, Ruffin MT, Brenner DE, Syngal S; Great Lakes-New England Clinical Epidemiology and Validation Center of the Early Detection Research Network. Missed adenomas during colonoscopic surveillance in individuals with Lynch Syndrome (hereditary nonpolyposis colorectal cancer). Cancer Prev Res (Phila). 2008 Nov;1(6):470-5. doi: 10.1158/1940-6207.CAPR-08-0098. PMID 19138994
- [Background] Huneburg R, Lammert F, Rabe C, Rahner N, Kahl P, Buttner R, Propping P, Sauerbruch T, Lamberti C. Chromocolonoscopy detects more adenomas than white light colonoscopy or narrow band imaging colonoscopy in hereditary nonpolyposis colorectal cancer screening. Endoscopy. 2009 Apr;41(4):316-22. doi: 10.1055/s-0028-1119628. Epub 2009 Apr 1. PMID 19340735
- [Background] Rahmi G, Lecomte T, Malka D, Maniere T, Le Rhun M, Guimbaud R, Lapalus MG, Le Sidaner A, Moussata D, Caron O, Barbieux JP, Gaudric M, Coron E, Barange K, Ponchon T, Sautereau D, Samaha E, Saurin JC, Chaussade S, Laurent-Puig P, Chatellier G, Cellier C. Impact of chromoscopy on adenoma detection in patients with Lynch syndrome: a prospective, multicenter, blinded, tandem colonoscopy study. Am J Gastroenterol. 2015 Feb;110(2):288-98. doi: 10.1038/ajg.2014.423. Epub 2015 Jan 20. PMID 25601014
- [Background] Rondagh EJ, Gulikers S, Gomez-Garcia EB, Vanlingen Y, Detisch Y, Winkens B, Vasen HF, Masclee AA, Sanduleanu S. Nonpolypoid colorectal neoplasms: a challenge in endoscopic surveillance of patients with Lynch syndrome. Endoscopy. 2013;45(4):257-64. doi: 10.1055/s-0032-1326195. Epub 2013 Feb 25. PMID 23440588
- [Background] Jass JR, Stewart SM. Evolution of hereditary non-polyposis colorectal cancer. Gut. 1992 Jun;33(6):783-6. doi: 10.1136/gut.33.6.783. PMID 1624160
- [Background] Rijcken FE, Hollema H, Kleibeuker JH. Proximal adenomas in hereditary non-polyposis colorectal cancer are prone to rapid malignant transformation. Gut. 2002 Mar;50(3):382-6. doi: 10.1136/gut.50.3.382. PMID 11839719
- [Background] Lindgren G, Liljegren A, Jaramillo E, Rubio C, Lindblom A. Adenoma prevalence and cancer risk in familial non-polyposis colorectal cancer. Gut. 2002 Feb;50(2):228-34. doi: 10.1136/gut.50.2.228. PMID 11788565
- [Background] Moller P, Seppala T, Bernstein I, Holinski-Feder E, Sala P, Evans DG, Lindblom A, Macrae F, Blanco I, Sijmons R, Jeffries J, Vasen H, Burn J, Nakken S, Hovig E, Rodland EA, Tharmaratnam K, de Vos Tot Nederveen Cappel WH, Hill J, Wijnen J, Green K, Lalloo F, Sunde L, Mints M, Bertario L, Pineda M, Navarro M, Morak M, Renkonen-Sinisalo L, Frayling IM, Plazzer JP, Pylvanainen K, Sampson JR, Capella G, Mecklin JP, Moslein G; Mallorca Group (http://mallorca-group.eu). Cancer incidence and survival in Lynch syndrome patients receiving colonoscopic and gynaecological surveillance: first report from the prospective Lynch syndrome database. Gut. 2017 Mar;66(3):464-472. doi: 10.1136/gutjnl-2015-309675. Epub 2015 Dec 9. PMID 26657901
- [Background] Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, Lehman GA, Mark DG. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies. Gastroenterology. 1997 Jan;112(1):24-8. doi: 10.1016/s0016-5085(97)70214-2. PMID 8978338
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Stoffel EM, Mangu PB, Gruber SB, Hamilton SR, Kalady MF, Lau MW, Lu KH, Roach N, Limburg PJ; American Society of Clinical Oncology; European Society of Clinical Oncology. Hereditary colorectal cancer syndromes: American Society of Clinical Oncology Clinical Practice Guideline endorsement of the familial risk-colorectal cancer: European Society for Medical Oncology Clinical Practice Guidelines. J Clin Oncol. 2015 Jan 10;33(2):209-17. doi: 10.1200/JCO.2014.58.1322. Epub 2014 Dec 1. PMID 25452455
- [Background] Balmana J, Balaguer F, Cervantes A, Arnold D; ESMO Guidelines Working Group. Familial risk-colorectal cancer: ESMO Clinical Practice Guidelines. Ann Oncol. 2013 Oct;24 Suppl 6:vi73-80. doi: 10.1093/annonc/mdt209. Epub 2013 Jun 27. No abstract available. PMID 23813931
- [Background] Vasen HF, Abdirahman M, Brohet R, Langers AM, Kleibeuker JH, van Kouwen M, Koornstra JJ, Boot H, Cats A, Dekker E, Sanduleanu S, Poley JW, Hardwick JC, de Vos Tot Nederveen Cappel WH, van der Meulen-de Jong AE, Tan TG, Jacobs MA, Mohamed FL, de Boer SY, van de Meeberg PC, Verhulst ML, Salemans JM, van Bentem N, Westerveld BD, Vecht J, Nagengast FM. One to 2-year surveillance intervals reduce risk of colorectal cancer in families with Lynch syndrome. Gastroenterology. 2010 Jun;138(7):2300-6. doi: 10.1053/j.gastro.2010.02.053. Epub 2010 Mar 2. PMID 20206180
- [Background] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Background] Chen SC, Rex DK. Endoscopist can be more powerful than age and male gender in predicting adenoma detection at colonoscopy. Am J Gastroenterol. 2007 Apr;102(4):856-61. doi: 10.1111/j.1572-0241.2006.01054.x. Epub 2007 Jan 11. PMID 17222317
- [Background] Kahi CJ, Hewett DG, Norton DL, Eckert GJ, Rex DK. Prevalence and variable detection of proximal colon serrated polyps during screening colonoscopy. Clin Gastroenterol Hepatol. 2011 Jan;9(1):42-6. doi: 10.1016/j.cgh.2010.09.013. Epub 2010 Oct 1. PMID 20888435
- [Background] Hazewinkel Y, Lopez-Ceron M, East JE, Rastogi A, Pellise M, Nakajima T, van Eeden S, Tytgat KM, Fockens P, Dekker E. Endoscopic features of sessile serrated adenomas: validation by international experts using high-resolution white-light endoscopy and narrow-band imaging. Gastrointest Endosc. 2013 Jun;77(6):916-24. doi: 10.1016/j.gie.2012.12.018. Epub 2013 Feb 21. PMID 23433877
- [Background] Kahi CJ, Li X, Eckert GJ, Rex DK. High colonoscopic prevalence of proximal colon serrated polyps in average-risk men and women. Gastrointest Endosc. 2012 Mar;75(3):515-20. doi: 10.1016/j.gie.2011.08.021. Epub 2011 Oct 21. PMID 22018551
- [Derived] Rivero-Sanchez L, Arnau-Collell C, Herrero J, Remedios D, Cubiella J, Garcia-Cougil M, Alvarez V, Albeniz E, Calvo P, Gordillo J, Puig I, Lopez-Vicente J, Huerta A, Lopez-Ceron M, Salces I, Penas B, Parejo S, Rodriguez de Santiago E, Herraiz M, Carretero C, Gimeno-Garcia AZ, Saperas E, Alvarez-Urturi C, Moreira R, Rodriguez de Miguel C, Ocana T, Moreira L, Carballal S, Sanchez A, Jung G, Castells A, Llach J, Balaguer F, Pellise M; EndoCAR group from Spanish Gastroenterology Association (AEG) and Spanish Society of Digestive Endoscopy (SEED). White-Light Endoscopy Is Adequate for Lynch Syndrome Surveillance in a Randomized and Noninferiority Study. Gastroenterology. 2020 Mar;158(4):895-904.e1. doi: 10.1053/j.gastro.2019.09.003. Epub 2019 Sep 12. PMID 31520613